CLINICAL TRIAL: NCT06436300
Title: Increasing Colorectal Cancer Screening in Alaska Native Men
Brief Title: Colorectal Cancer Screening in Alaska Native Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: Southcentral Foundation (Other)
Responsible Party: Principal Investigator, Clemma Muller, Associate Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: R21NR019362 (NIH)
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
Keywords: screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel arm randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Usual care arm receives established methods for scheduling colorectal cancer screening with clinic patients.
- Messages only (Experimental): Receives motivational messages to promote colorectal cancer screening plus usual care.
  Interventions: Behavioral: Motivational text messaging
- Messages plus gift card (Experimental): Receives motivational messages to promote colorectal cancer screening, plus offer of a $50 gift card for completing screening, plus usual care.
  Interventions: Behavioral: Motivational text messaging
- Messages plus raffle (Experimental): Receives motivational messages to promote colorectal cancer screening, plus offer of entry into a raffle for a prize worth approximately $200 if they complete screening, plus usual care.
  Interventions: Behavioral: Motivational text messaging

INTERVENTIONS:
Behavioral: Motivational text messaging — Intervention sends up to 4 motivational messages by text or email to Alaska Native men who are active patients and due for colorectal cancer screening. Incentive arms include promise of a $50 gift card or entry into a raffle for prize worth about $200 if they complete screening.
  Arms: Messages only; Messages plus gift card; Messages plus raffle

SUMMARY:
Alaska Native men have the highest rates of colorectal cancer incidence and mortality in the US. Screening can prevent disease and improve survival. A previous study tested text messages to increase colorectal cancer screening in Alaska Native patients of the Southcentral Foundation healthcare system in Anchorage, Alaska. The intervention improved screening by 50% in women, but it had no effect in men. The current study aimed to culturally tailor the intervention for Alaska Native Men, and to test it with a randomized controlled trial among patients at the Southcentral Foundation.

DETAILED DESCRIPTION:
Alaska Native men have higher colorectal cancer (CRC) incidence and mortality than any other US racial or ethnic group. Screening can prevent CRC and improve treatment outcomes by detecting disease in early stages, but Alaska Native men also have low CRC screening uptake. Colonoscopy is the most accurate CRC screening method and results in the most years of life saved. It only requires rescreening every 10 years, but it is a clinic- based procedure and needs extensive preparation. Other screening options include home-based tests that detect blood in the stool and require rescreening every year. More recently, a home-based method has been developed that tests stool for DNA indicative of CRC and requires rescreening every 3 years. Current guidelines recommend CRC screening for average risk adults starting between ages 45-50, but people at higher risk should start at younger ages. Many interventions have been developed to promote CRC screening. Among these, interventions that use text messaging or other electronic health messages to reach people outside of the clinical setting have shown promise for improving CRC screening. In a previous study, the research team developed an intervention that sends up to 3 text messages to Alaska Native people patients of the Southcentral Foundation (SCF) healthcare system in Anchorage, Alaska. The intervention was tested in a randomized controlled trial with 2,386 Alaska Native SCF patients ages 40-75. The intervention increased CRC screening by 50% in women, but it had no effect in men. The current study used a theory-based approach to culturally tailor the previous text message intervention for Alaska Native men. Investigators conducted a randomized trial to test the effectiveness of the tailored intervention with 998 Alaska Native men ages 40-75 who were active patients at SCF. Eligible men were identified from the electronic medical record and randomized in equal proportions to the control condition or to one of three intervention arms (messages only, messages plus gift card incentive, messages plus raffle incentive). The primary outcomes were completed CRC screening documented in the electronic medical record within 6 months of sending the first text message, and any scheduled visit for pre-screening or screening documented in the medical record during follow-up. The study obtained a waiver of consent, and no individuals were directly recruited or enrolled in the study. Follow-up was entirely ascertained through the electronic medical record, and cohort attrition was not applicable.

ELIGIBILITY:
Inclusion Criteria:

* Alaska Native or American Indian racial identity
* Male gender identity
* Active patient of the Southcentral Foundation in Anchorage, Alaska
* Empanelled to primary care provider in the Anchorage or local Valley area
* Eligible for routine preventive colorectal cancer screening

Exclusion Criteria:

* None

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility determined in the electronic medical record, which reflects gender identity.
Enrollment: 998 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Southcentral Foundation, Anchorage, Alaska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial obtained a waiver of consent, and no individuals were directly recruited or enrolled. Screening-eligible men who met all other criteria were identified in the electronic health record and randomly sampled for inclusion in the study cohort.
Pre-assignment Details: Prior to sending the first electronic message, we re-queried the electronic health record and removed men who had completed colorectal screening in the interval between randomization and launching the trial.
Groups:
- Control: The control arm received usual care for colorectal cancer screening outreach, and did not receive any study-related electronic messages.
- Messages: This arm received electronic messages to promote colorectal cancer screening, but did not receive any notices about additional incentives.
- Gift Card: This arm received the same electronic messages as the "Messages" arm, and was additionally promised a $50 gift card if they completed colorectal screening by the target date.
- Raffle: This arm received the same electronic messages as the "Messages" arm, and were additionally promised they would be added to a raffle (~$200 prize value) if they completed screening before a target date.
Period: Overall Study
Arm/Group | Control | Messages | Gift Card | Raffle
Started | 250 | 250 | 248 | 250
Completed (The outcome was colorectal cancer screening documented in the electronic health record, which enabled 100% follow-up.) | 250 | 250 | 248 | 250
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Messages | Gift Card | Raffle | Total
Number analyzed (Participants) | 250 | 250 | 248 | 250 | 998
Sex: Female, Male [Count of Participants; unit: Participants] — This study only included patients identified as male in the electronic health record
  Participants
    Female | 0 | 0 | 0 | 0 | 0
    Male | 250 | 250 | 248 | 250 | 998
Race (NIH/OMB) [Count of Participants; unit: Participants] — This study only included men identified as Alaska Native or American Indian in the electronic health record.
  Participants
    American Indian or Alaska Native | 250 | 250 | 248 | 250 | 998
    Asian | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Previous screening [Count of Participants; unit: Participants] — Any previous colorectal cancer screening documented in the electronic health record
  Participants
    Previously screened | 36 | 40 | 36 | 40 | 152
    Not previously screened | 214 | 210 | 212 | 210 | 846
Age, Customized [Count of Participants; unit: Participants]
  40-44 years | 78 | 82 | 87 | 79 | 326
  45-49 years | 47 | 47 | 40 | 47 | 181
  50-54 years | 46 | 40 | 39 | 29 | 154
  55-59 years | 29 | 29 | 26 | 32 | 116
  60-65 years | 50 | 52 | 56 | 63 | 221

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed Colorectal Cancer Screening
Description: Screening procedure documented in the electronic medical record
Time Frame: Six months
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Messages | Gift Card | Raffle
Number analyzed (Participants) | 250 | 250 | 248 | 250
Participants
  Any screening documented | 11 | 16 | 18 | 19
  No screening documented | 239 | 234 | 230 | 231

2. Primary Outcome: Number of Participants Who Scheduled a Screening-related Visit
Description: Pre-screening or screening visit scheduled in the electronic medical record during follow-up
Time Frame: Six months
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Messages | Gift Card | Raffle
Number analyzed (Participants) | 250 | 250 | 248 | 250
Participants
  Visit scheduled | 8 | 20 | 18 | 17
  No visit scheduled | 242 | 230 | 230 | 233

ADVERSE EVENTS:
Time Frame: Six months, from date of randomization to end of follow-up
Arm/Group | Control | Messages | Gift Card | Raffle
All-Cause Mortality (participants affected / at risk) | 0/250 | 0/250 | 0/248 | 0/250
Serious Adverse Events (participants affected / at risk) | 0/250 | 0/250 | 0/248 | 0/250
Other Adverse Events (participants affected / at risk) | 0/250 | 0/250 | 0/248 | 0/250

LIMITATIONS AND CAVEATS:
This study was limited to male patients at a single Tribal health care system in the Anchorage Metropolitan Area. Results may not generalize to other Alaska Native or American Indian people in other locations or settings.

Colorectal cancer screening performed outside of the health care system would not be included in outcome data, but the vast majority of patients receive most or all their care from the Southcentral Foundation and we anticipate minimial misclassification of screening.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT06436300/Prot_SAP_000.pdf